CLINICAL TRIAL: NCT01900639
Title: Effect of Aspirin Intake on Awakening Versus at Bedtime on Circadian Rhythm of Platelet Reactivity in Healthy Subjects
Brief Title: Aspirin AM or PM: Effect on Circadian Rhythm of Platelet Reactivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NL.44378.058.13; 2013-001410-16 (EudraCT Number); P13.092 (Other: Leiden University Medical Center)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Aspirin; Circadian Rhythm; Platelet Activation; Cardiovascular Diseases
Keywords: aspirin; circadian rhythm; platelet reactivity; platelet activation; time dependent
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aspirin on awakening (Active Comparator): intake of 80 acetylsalicylic acid on awakening for 2 weeks
  Interventions: Behavioral: change time of intake of aspirin
- aspirin at bedtime (Experimental): intake of 80mg acetylsalicylic acis at bedtime
  Interventions: Behavioral: change time of intake of aspirin

INTERVENTIONS:
Behavioral: change time of intake of aspirin

SUMMARY:
Low-dose aspirin is a cornerstone in the secondary prevention of cardiovascular disease (CVD) and is usually taken on awakening, although evidence regarding optimal time of intake is lacking. Platelet reactivity follows a circadian rhythm, with a peak in the morning, contributing to the morning peak of cardiovascular disease. Due to its short half life, aspirin only inhibits platelets which are present at the time of intake. Thus, the timing of aspirin intake may influence its inhibitory effect on platelets and intake of aspirin at bedtime may attenuate the morning peak of platelet reactivity. The time-dependent effect of aspirin on circadian rhythm of platelet function has never been studied before. We hypothesize that aspirin intake at bedtime compared with intake on awakening results in a reduction of the morning peak in platelet reactivity.

DETAILED DESCRIPTION:
Cardiovascular events are a leading cause of mortality and morbidity in western countries. In the European Union, 47% of total mortality is caused by cardiovascular disease2. Aspirin is a cornerstone in the secondary prevention of cardiovascular disease because of its inhibitory effects on platelet aggregation. It reduces the risk of recurrent cardiovascular events with about a quarter3. Although not supported by evidence, aspirin is usually taken in the morning, but it may be more beneficial to take aspirin at bedtime instead of on awakening. It has been convincingly shown that platelet activity follows a circadian rhythm, with a peak of platelet reactivity in the morning4-8. This might in part explain the increase in cardiovascular events in the early morning, with the highest incidence between 6 and 12 AM1.

Since platelet reactivity follows a circadian rhythm, the timing of aspirin intake may influence its inhibitory effect on platelets. Due to its short half-life, aspirin only inhibits platelets which are present at the time of intake. New platelets are released at a rate of 10%/day, predominantly during the night9. Because they are more reactive and not inhibited by aspirin taken in the preceding morning, these young platelets contribute to the morning peak of platelet reactivity10, 11. It has been argued that intake of aspirin at bedtime could better prevent the early morning increase in platelet reactivity than intake on awakening, assuming that intake on awakening would be too late to prevent this morning peak in platelet reactivity12. Additionally, a recent study showed significant recovery of platelet aggregation after 24 hours in patients using low-dose aspirin on a daily basis13. This supports the hypothesis that aspirin intake at bedtime could be beneficial in reducing the morning peak of platelet reactivity, thereby possibly also reducing the incidence of arterial thrombotic events in the morning. However, this has never been studied before.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Age >18yrs
* Capacity to give informed consent (IC)

Exclusion Criteria:

* Active chronic disease
* Use of any other medication
* History of: major bleeding events, known bleeding diathesis or disorder, cardiovascular disease, malignancy
* Known allergy to salicylates
* Platelet count < 150 * 109/L
* VerifyNow Aspirin Reaction Units <550 Aspirin Reaction Units (ARU)
* Smoking
* Shift work in preceding 2 months
* Extreme chronotypes, defined as regular (>2 days/week) bedtime <22:00h or >24:00h and/or awakening <6:00h or >9:00h
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm of platelet reactivity | 24hour rhythm of platelet reactivity
  Platelet reactivity will be measured by VerifyNow-aspirin assay, serum thromboxane B2, and flow-cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Tofler GH, Brezinski D, Schafer AI, Czeisler CA, Rutherford JD, Willich SN, Gleason RE, Williams GH, Muller JE. Concurrent morning increase in platelet aggregability and the risk of myocardial infarction and sudden cardiac death. N Engl J Med. 1987 Jun 11;316(24):1514-8. doi: 10.1056/NEJM198706113162405. PMID 3587281
- [Background] Scheer FA, Michelson AD, Frelinger AL 3rd, Evoniuk H, Kelly EE, McCarthy M, Doamekpor LA, Barnard MR, Shea SA. The human endogenous circadian system causes greatest platelet activation during the biological morning independent of behaviors. PLoS One. 2011;6(9):e24549. doi: 10.1371/journal.pone.0024549. Epub 2011 Sep 8. PMID 21931750
- [Background] Di Minno G, Silver MJ, Murphy S. Monitoring the entry of new platelets into the circulation after ingestion of aspirin. Blood. 1983 Jun;61(6):1081-5. PMID 6404326
- [Background] Kriszbacher I, Ajtay Z, Koppan M, Bodis J. Can the time of taking aspirin influence the frequency of cardiovascular events? Am J Cardiol. 2005 Aug 15;96(4):608-10. doi: 10.1016/j.amjcard.2005.03.068. No abstract available. PMID 16098324
- [Derived] Bonten TN, Saris A, van Oostrom MJ, Snoep JD, Rosendaal FR, Zwaginga J, Eikenboom J, van der Meer PF, van der Bom JG. Effect of aspirin intake at bedtime versus on awakening on circadian rhythm of platelet reactivity. A randomised cross-over trial. Thromb Haemost. 2014 Dec;112(6):1209-18. doi: 10.1160/TH14-05-0453. Epub 2014 Sep 11. PMID 25208590